CLINICAL TRIAL: NCT07368712
Title: Study to Investigate Renal Functional Reserve in Healthy Participants and in Participants With Impaired Renal Function.
Brief Title: A Methodological Study to Learn More About Kidney Function in Healthy People and in People With Reduced Kidney Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23125
Record Dates: First submitted 2026-01-02; First posted 2026-01-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Kidney Injury, Renal Insufficiency
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other)
  Interventions: Other: No investigational study intervention

INTERVENTIONS:
Other: No investigational study intervention — The study does not involve the administration of any study intervention, investigational medicinal product, or device. Participants will undergo blood collection and urine sampling both before and after consuming a high-protein meal.

SUMMARY:
The main purpose of this study is to investigate how reliable a test assessing the renal functional reserve (RFR) and the maximum glomerular filtration rate (maxGFR) are. MaxGFR and RFR assessments are repeated twice at 1-month intervals. If precise, this test may improve the measure of kidney function and be useful in future studies for people with chronic kidney problems.

To do this, the researchers will collect and analyze information about kidney function from up to 50 adults, including healthy people and people with stable kidney problems. Each person will come to the study center for a screening visit and then three study days, each about a month apart. On each study day, participants will have blood and urine samples taken before and after drinking a protein shake. The tests will measure things like creatinine, cystatin C, and other markers in the blood and urine to see how the kidneys are working. The study will also record basic health information, weight, blood pressure, and any medicines being taken.

The study will last about 2 to 2.5 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 75 years of age inclusive, at the time of signing the ICF.
* Stable medical condition defined as no new drug or other treatment prescribed for a chronic condition within 60 days prior to Study Day 1.
* Body weight between 50 and 100 kg.
* Female Participants: A participant is eligible to participate if not pregnant or breastfeeding. If a urine test cannot be confirmed as negative at screening (e.g., an ambiguous result), the participant must be excluded from participation.

Exclusion Criteria:

* Recent surgical intervention within 60 days prior to Study Day 1.
* New clinical diagnosis established within 60 days prior to Study Day 1.
* New drug prescription within 60 days prior to Study Day 1.
* Relevant change in severity of any medical condition within 60 days prior to Study Day 1, e.g. disease flare.
* Known congenital amino acid metabolism disorders.
* Severe hypersensitivity to milk products.
* Known liver cirrhosis.
* Regular use of non-steroidal anti-inflammatory drugs (NSAIDs).
* Impaired kidney function with eGFR <30 mL/min/1.73m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Maximun kidneyfunction determined by measurement of creatinine clearance (mGFRCR) | Day 1, 28 and 56
Renal functional reserve by measurement of creatinine clearance (mGFRCR) | Day 1, 28 and 56

SECONDARY OUTCOMES:
Maximum kidney function and renal functional reserve derived from serum creatinine-based eGFR (eGFRSCR) | Day 1, 28 and 56
Maximum kidney function and renal functional reserve derived from serum cystatin C-based eGFR (eGFRCYS) | Day 1, 28 and 56
Maximum kidney function and renal functional reserve derived from serum creatinine-based and serum cystatin C-based eGFR (eGFRSCR-CYS) | Day 1, 28 and 56
Maximum creatinine clearance and renal functional reserve derived from plasma PENK-based eGFR (eGFRPENK) | Day 1, 28 and 56

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer AG - Occupational Health Services, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access. As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.